CLINICAL TRIAL: NCT00450996
Title: Phase 3: Analysis of a Beneficial Effect of Prolonges Topical Steroid Treatment After Low-risk Penetrating Keratoplasty
Brief Title: Analysis of a Beneficial Effect of Prolonges Topical Steroid Treatment After Low-risk Penetrating Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PostkeratoplastySteroids
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Graft Rejection
MeSH Terms: interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topical Steroids

SUMMARY:
PURPOSE: To assess the impact of duration of topical steroid treatment on the incidence of endothelial graft rejection following normal-risk penetrating keratoplasty (PK). DESIGN: Prospective, institutional, longitudinal, randomized interventional trial including 406 eyes (age: 52 >= 19 years; follow-up: 42 >= 18months). METHODS: Postoperative treatment started with prednisolone acetate 1% eye drops five times daily and was tapered over the first 6 months. Patients were then randomised into either short-term (stop topical steroid treatment) or long-term treatment (continue steroids once daily until 12 months).

DETAILED DESCRIPTION:
PURPOSE: To assess the impact of duration of topical steroid treatment on the incidence of endothelial graft rejection following normal-risk penetrating keratoplasty (PK). DESIGN: Prospective, institutional, longitudinal, randomized interventional trial including 406 eyes (age: 52 >= 19 years; follow-up: 42 >= 18 months). METHODS: Postoperative treatment started with prednisolone acetate 1% eye drops five times daily and was tapered over the first 6 months. Patients were then randomised into either short-term (stop topical steroid treatment) or long-term treatment (continue steroids once daily until 12 months). <=

ELIGIBILITY:
Inclusion Criteria:

* Low risk keratoplasty

Exclusion Criteria:

* High risk keratoplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1999-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Graft survival

CONTACTS AND LOCATIONS:
Overall Officials: friedrich Naumann, MD, Principal Investigator — University of Erlangen-Nürnberg; claus Cursiefen, md, Study Director — University of Erlangen-Nürnberg